CLINICAL TRIAL: NCT00609336
Title: A Phase II Study Induction Chemotherapy, Neoadjuvant Chemoradiotherapy, Surgical Resection and Adjuvant Chemotherapy for Patients With Locally Advanced, Resectable Pancreatic Adenocarcinoma
Brief Title: Perioperative Therapy for Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Coveler, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6511; NCI-2010-00553 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6511 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-07 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Adenocarcinoma of the Pancreas; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine; Radiotherapy, Intensity-Modulated; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, radiation, pancreaticoduodenectomy) (Experimental): See Detailed Description
  Interventions: Drug: gemcitabine hydrochloride; Drug: docetaxel; Drug: capecitabine; Radiation: intensity-modulated radiation therapy; Drug: oxaliplatin; Procedure: pancreatic surgical procedure; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Radiation: intensity-modulated radiation therapy — Undergo IMRT
  Other Names: IMRT
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Procedure: pancreatic surgical procedure — Undergo pancreaticoduodenectomy
  Other Names: pancreatic surgery
Procedure: therapeutic conventional surgery — Undergo therapeutic conventional surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving combination chemotherapy together with intensity-modulated radiation therapy (IMRT) and surgery works in treating patients with localized pancreatic cancer that can be removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride, docetaxel, capecitabine, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Specialized radiation therapy, such as IMRT, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving more than one drug (combination chemotherapy) together with intensity-modulated radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the median overall survival of patients with adenocarcinoma of the pancreas treated with induction chemotherapy, neoadjuvant chemoradiotherapy, surgical resection and adjuvant chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the percent of patients surviving at annual intervals through five years.

II. To determine the median recurrence free survival following pancreaticoduodenectomy.

III. To determine the clinical response rate to neoadjuvant chemotherapy and chemoradiotherapy.

IV. To determine the pathologic response rate to neoadjuvant chemotherapy and chemoradiotherapy.

V. To determine the cancer antigen (CA) 19-9 tumor marker response rate to neoadjuvant chemotherapy and chemoradiotherapy.

VI. To determine the surgical completion rate and complication rate following neoadjuvant chemotherapy and chemoradiotherapy.

VII. To determine the frequency and severity of toxicities associated with this treatment regimen.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive gemcitabine hydrochloride intravenously (IV) over 75 minutes and docetaxel IV over 30 or 60 minutes on days 4 and 11. Patients also receive capecitabine orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

NEOADJUVANT CHEMORADIOTHERAPY: Beginning no more than 14 days after completion of induction chemotherapy, patients receive capecitabine PO BID on days 1-14 and oxaliplatin IV over 2 hours on days 1 and 8. Patients also undergo IMRT once daily on days 1-5 and 8-13.

SURGICAL RESECTION: Approximately 2-6 weeks after completion of neoadjuvant chemoradiotherapy, patients undergo pancreaticoduodenectomy.

ADJUVANT CHEMOTHERAPY: Beginning 4-10 weeks after surgery, patients receive gemcitabine hydrochloride IV over 30 minutes and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients then receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of localized, resectable or borderline resectable, pancreatic adenocarcinoma T1-T3, N0-N1, M0; stage is determined by helical multi-phase computed tomography (CT) and/or endoscopic ultrasound according to published guidelines; resectability is determined by the treating surgeon and published guidelines (National Comprehensive Cancer Network)
* Resectable Disease- Head/Body/Tail of pancreas:

  * No distant metastases
  * Clear fat plane around celiac and superior mesenteric arteries (SMA)
  * Patent superior mesenteric vein (SMV) and portal vein (PV)
* Borderline Resectable Disease -Head/Body of pancreas:

  * Tumor abutment on SMA
  * SMV/portal vein impingement or occlusion if involving only a short segment, with open vein both proximally and distally (if proximal vein is occluded up to the portal vein branches then disease is unresectable)
  * Colon or mesocolon invasion
  * Gastroduodenal artery (GDA) encasement up to origin at hepatic artery
* Tail of pancreas:

  * Adrenal, colon or mesocolon, or kidney invasion
  * Preoperative evidence of biopsy-positive peripancreatic lymph node
* No prior therapy for pancreatic cancer
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leucocytes >= 3,000/uL
* Absolute Neutrophil Count >= 1,500/uL
* Platelets >= 100,000/uL
* Total Bilirubin:

  * If within normal limits (WNL) to =< 2.0, the subject is eligible
  * If > 2.0 - < 6.0, subject is eligible IF they have a biliary stent and total bilirubin is decreasing
  * If >= 6.0, subject is not eligible
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal or =< 1.5 X upper limit of normal (ULN) if alkaline phosphatase (Alk Phos) > 2.5 X ULN or if the subject has a biliary stent and the liver function tests (LFTs) are decreasing the subject is eligible
* Creatinine clearance >= 30%
* Negative pregnancy test for women of childbearing potential; women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to swallow and retain oral medication
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Histology other than adenocarcinoma
* Patients with permanently unresectable pancreatic adenocarcinoma as determined by the treating physician and published guidelines (National Comprehensive Cancer Network)
* Unresectable disease
* Head of pancreas:

  * Distant metastases (includes celiac and/or para-aortic)
  * SMA, celiac encasement
  * SMV/portal occlusion
  * Aortic, inferior vena cava (IVC) invasion or encasement
  * Invasion of SMV below transverse mesocolon
* Body of pancreas:

  * Distant metastases (includes celiac and/or para-aortic); at the discretion of the treating surgeon, body and tail lesions that have positive celiac and/or para-aortic nodes in close vicinity to the primary may be borderline rather than unresectable
  * SMA, celiac, hepatic encasement
  * SMV/portal extended occlusion
  * Aortic invasion
* Tail of pancreas:

  * Distant metastases (includes celiac and/or para-aortic)
  * SMA, celiac encasement
  * Rib, vertebral invasion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, docetaxel, capecitabine, oxaliplatin or other agents used in the study
* Patients who have received prior chemotherapy or radiotherapy for the diagnosis of pancreatic cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Inability to comply with study and/or follow-up procedures
* Pregnancy or lactation
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2014-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Coveler, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy): See Detailed Description
  gemcitabine hydrochloride: Given IV
  docetaxel: Given IV
  capecitabine: Given PO
  intensity-modulated radiation therapy: Undergo IMRT
  oxaliplatin: Given IV
  pancreatic surgical procedure: Undergo pancreaticoduodenectomy
  therapeutic conventional surgery: Undergo therapeutic conventional surgery
  gemcitabine: Given IV
  oxaliplatin: Given IV
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Started | 35
Surgery | 22
Completed | 22
Not Completed | 13
Not completed — Protocol Violation | 3
Not completed — Death | 1
Not completed — LA or Met at Surgery | 9

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival of Patients With Adenocarcinoma of the Pancreas
Description: Time at which Kaplan-Meier estimate of overall survival drops below 50%
Time Frame: 5 years
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 32
months | 31.6 [14.2 to 58.1]

2. Secondary Outcome: Percent of Patients Surviving at 5 Years
Description: Kaplan-Meier estimate of overall survival at 5 years
Time Frame: Up to 5 years
Population: all eligible patients
Measure: Number; unit: percentage of eligible pts alive
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 32
percentage of eligible pts alive | 31.6

3. Secondary Outcome: Median Recurrence Free Survival Following Pancreaticoduodenectomy
Description: The appearance of radiographic findings consistent with recurrent tumor at the local resection site or at a distant location is considered a radiographic recurrence.
Time Frame: From the date of pancreaticoduodenectomy to date of first observation of radiographic recurrence or death due to any cause, assessed up to 7 years
Population: Among eligible patients who received surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 22
months | 31.3 [12.5 to NA] — Upper limit is infinite.

4. Secondary Outcome: Clinical Response Rate to Neoadjuvant Chemotherapy and Chemoradiotherapy
Description: Assessed using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.
Time Frame: Up to 7 years
Population: Clinical response not collected.
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Pathologic Response Rate (Complete, Near-complete, Partial) to Neoadjuvant Chemotherapy and Chemoradiotherapy
Description: The resected pancreaticoduodenectomy specimen and accompanying lymph nodes will be staged according to American Joint Committee on Cancer 6th Edition incorporating the prefix y to indicate a specimen status-post neoadjuvant treatment (ypTNM). Cancer 2012;118:1382-90
Time Frame: Up to 7 years
Population: all eligible patients with non-missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 22
Participants | 20

6. Secondary Outcome: CA 19-9 Tumor Marker Response Rate to Neoadjuvant Chemotherapy and Chemoradiotherapy
Description: Biochemical response is a decrease of >= 50% of CA 19-9 serum tumor marker in patients with elevated CA 19-9 at baseline.
Time Frame: Up to 26 weeks after surgery
Population: Biomarker data not collected.
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Surgical Completion Rate and Complication Rate
Time Frame: Up to 6 weeks following the completion of chemoradiotherapy
Population: all eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 32
Participants
  Completion rate | 22
  Complication rate: number analyzed (Participants) | 22
  Complication rate | 2

8. Secondary Outcome: Frequency and Severity of Toxicities Associated With This Treatment Regimen as Assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: Up to 26 weeks after surgery (the end of adjuvant chemotherapy)
Population: All eligible patients
Measure: Number; unit: occurrence of toxicities
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 32
occurrence of toxicities
  Any Grade 2 CTCAE toxicity | 21
  Any Grade 3 CTCAE toxicity | 121
  Any Grade 4 CTCAE toxicity | 14

9. Secondary Outcome: Percent of Patients Surviving at Annual Intervals
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Number analyzed (Participants) | 32
percentage of participants
  Year 1 | 81
  Year 2 | 62
  Year 3 | 45
  Year 4 | 37
  Year 5 | 31

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy)
Serious Adverse Events (participants affected / at risk) | 32/35
Other Adverse Events (participants affected / at risk) | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy) (N=35)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Elevated Bilirubin (Investigations) | 4 (4)
Fever, Neutropenic (Blood and lymphatic system disorders) | 3 (3)
Hand-foot Syndrome (Skin and subcutaneous tissue disorders) | 20 (22)
Infection (Infections and infestations) | 1 (2)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 24 (31)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (12)
Vomiting (Gastrointestinal disorders) | 2 (2)
Anasarca (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholangitis With Stent Occlusion (Hepatobiliary disorders) | 1 (1)
Cholecystic Abcess (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Entero Cutaneous Fistula (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Hypertension (Vascular disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoatremic (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Intrahepatic Absesses (Hepatobiliary disorders) | 1 (1)
Lower GI Bleed (Gastrointestinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (2)
Non-Malignant Ascitess (Hepatobiliary disorders) | 1 (1)
Nose Bleeds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive Jaundice (Hepatobiliary disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Shoulder Pain (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Transient Ischemic Attacks (Cardiac disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Radiation, Pancreaticoduodenectomy) (N=32)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 7 (8)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Elevated Bilirubin (Investigations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Maculopapular Rash (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash - Upper Torso (Skin and subcutaneous tissue disorders) | 1 (1)
Transaminase (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes